CLINICAL TRIAL: NCT03051750
Title: Complex Physical Therapy Plus Pressotherapy Versus Kinesio Taping in Breast Cancer-Related Lymphedema. Randomized Crossover Trial.
Brief Title: Comparison of Techniques for Breast Cancer-Related Lymphedema.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Violeta Pajero Otero (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other); University of Castilla-La Mancha (Other)
Responsible Party: Sponsor-Investigator, Violeta Pajero Otero, Physiotherapist at the Mammary Pathology Unit, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: InveCuidRh150316
Record Dates: First submitted 2017-02-08; First posted 2017-02-14 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer Lymphedema
Keywords: Breast Cancer-Related Lymphedema; Complex Physical Therapy; Pressotherapy; Kinesio Taping; Physiotherapy; Manual Lymph Drainage; Multilayer Bandage; TTDL questionnaire
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Intervention Model Description: 3-month previous washout period; 3-week treatment phases; 3-month washout period between both treatment phases.
  Open design: it is impossible during the treatment to blind the physiotherapists and patients, due to the observable differences between both therapies both during their application and in the hours after their removal, by the marks that leave in the skin.
  Interventions: The two therapies compared are:
  * CPT+ P.
  * KT.
Who Masked: Outcomes Assessor
Masking Description: The statistical analysis will be supervised by staff of the Scientific Support Unit: Epidemiology and Biostatistics (i+12), Hospital Universitario 12 de Octubre with the variables coded to blind the analyst.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPT+P (Active Comparator): Complex Physical Therapy plus Pressotherapy during three weeks
  Interventions: Other: Complex Physical Therapy plus Pressotherapy
- Kinesio Taping (Experimental): Kinesio Taping during three weeks
  Interventions: Other: Kinesio Taping

INTERVENTIONS:
Other: Complex Physical Therapy plus Pressotherapy
  Arms: CPT+P
Other: Kinesio Taping
  Arms: Kinesio Taping

SUMMARY:
This crossover study compares two different treatment techniques for Breast Cancer-Related Lymphedema: 1. Complex Physical Therapy plus Pressotherapy.

2. Kinesio Taping.

DETAILED DESCRIPTION:
Breast Cancer-Related Lymphedema (BCRL) tends to progress in stage and grade if it is not treated.

Complex Physical Therapy (CPT), that includes Manual Lymph Drainage + Multilayer Bandage + Self-care, is the most used technique in order to join the benefits of each technique by the lack of great results with only one technique. The most volume reduction found in a study was achieved combining CPT and Pressotherapy(P). On the other hand, the use of Kinesio Taping (KT) for BCRL has been spreading lately although its clinical efficacy has not been determined by high quality studies.

GOALS:

Main objective: To analyze the effectiveness in the reduction of BCRL volume with KT versus CPT+P in patients attended at the rehabilitation service at HU12Octubre.

Secondary objectives:

To analyze possible changes after each therapy in:

* DASH (Disability Arm, Shoulder and Hand) outcome measure score.
* TTDL (textile therapeutic device for lymphedema) questionnaire score (a quality of life questionnaire for patients with breast cancer-related upper lymb lymphedema using textile therapeutic device that has been validated previously).
* Symptoms associated with BCRL (pain, heaviness, pressure and hardness) using visual analogue scale (VAS).
* Goniometry of Upper Limb.

METHODOLOGY OF THE STUDY:

Design: crossover trial, with a 3-month washout period between both treatment phases. Open design: it is impossible during the treatment to blind physiotherapists and patients, due to the observable differences between both therapies neither during their application nor in the hours after their removal, by the marks left in the skin. The statistical analysis will be supervised by staff of the Clinical Research Unit-Clinical Trials (i+12) of HU12Octubre with the variables coded to blind the analyst.

Interventions: The two therapies compared are:

* CPT+ P.
* KT. Sample size: a sample of 50 patients (25 in each group) was calculated. Subjects of study and randomization: An initial computerized randomized sample was generated among the patients who had attended the Breast Pathology Rehabilitation visit at HU12Octubre during the previous year and who met the eligibility criteria and they were randomly assigned to the groups.

ELIGIBILITY:
Inclusion Criteria:

1. Submit BCRL
2. Be a patient of the Breast Pathology Rehabilitation at Hospital Universitario 12 de Octubre.
3. Signing the informed consent.

Exclusion Criteria:

1) Breast Cancer metastasis or other active tumor. 2) Intravenous chemotherapy or radiotherapy actually. 3) Heart or kidney failure. 4) Use diuretics. 5) active infection (erysipelas) or any cutaneous disease in UL or back. 5) Bilateral lymphadenectomy. 6) present deterioration or cognitive delay that would prevent understanding instructions and purpose of the study.

7) Have performed treatment for BCRL during the 3 months prior to the start of the study (previous washing phase).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 43 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Changes in the volume difference between the upper limb with lymphedema and the healthy upper limb before and after treatment. | Four weeks during each treatment phase
  Truncated Cone Formula for Volume from upper limb circumference.

SECONDARY OUTCOMES:
Score on the DASH Outcome Measure. | Four weeks during each treatment phase
  Validated questionnaire about Disability of the Arm,Shoulder and Hand.
Score of the TTDL questionnaire. | Four weeks during each treatment phase
  a quality of life questionnaire for patients with breast cancer-related upper lymphedema using textile therapeutic device validated previously (not yet published).
Symptoms associated with BCRL (pain, heaviness, pressure and hardness) using modified visual analogue scale (VAS). | Four weeks during each treatment phase
  Wong-Baker faces pain rating scale.
Stage of the lymphedema. | Four weeks during each treatment phase
  I, IIA, IIB III, IV.
Goniometry of Upper Limb. | Four weeks during each treatment phase
  Goniometry of shoulder, elbow and wrist.
Body Mass Index. | Four weeks during each treatment phase
  The weight in kilograms divided by the square of the height in metres (kg/m2).

OTHER OUTCOMES:
Age. | First day of treatment of the first phase.
  Years old at the beginning of the study.
Time since axillary surgery. | First day of treatment of the first phase.
  Time since axillary surgery in years at the beginning of the study.
Type of axillary surgery. | First day of treatment of the first phase.
  Lymphadenectomy or Sentinel Lymph Node Biopsy.
Type of breast surgery. | First day of treatment of the first phase.
  Lumpectomy or mastectomy.
Radiotherapy for Breast Cancer. | First day of treatment of the first phase.
  Yes or not.
Time since the appearance of the BCRL. | First day of treatment of the first phase.
  Years since the BCRL appeared.

CONTACTS AND LOCATIONS:
Overall Officials: Violeta Pajero Otero, MRes, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pajero Otero V, Garcia Delgado E, Martin Cortijo C, Rodriguez Ramos ML, De Carlos Iriarte E, Gil Garcia A, Romay-Barrero H, Avendano-Coy J. Intensive complex physical therapy combined with intermittent pneumatic compression versus Kinesio taping for treating breast cancer-related lymphedema of the upper limb: A randomised cross-over clinical trial. Eur J Cancer Care (Engl). 2022 Sep;31(5):e13625. doi: 10.1111/ecc.13625. Epub 2022 May 31. PMID 35642305